CLINICAL TRIAL: NCT02087644
Title: A Randomized, Placebo-Controlled, Phase IIb Study of CYT003-QbG10 (CYT003), a TLR9 Agonist, in Patients With Mild to Moderate Allergic Asthma Not Sufficiently Controlled on Inhaled Glucocorticosteroids
Brief Title: CYT003 in Patients With Mild to Moderate Allergic Asthma Not Sufficiently Controlled on Inhaled Glucocorticosteroids
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT003-QbG10 13
Record Dates: First submitted 2014-03-11; First posted 2014-03-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — CYT003-QbG10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYT003 (Experimental): Injections of CYT003
  Interventions: Biological: CYT003
- Placebo (Placebo Comparator): Injections of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CYT003 — Injections
  Arms: CYT003
Biological: Placebo — Injections
  Arms: Placebo

SUMMARY:
A phase IIb study in patients to evaluate CYT003- QbG10 versus placebo, in patients with mild to moderate allergic asthma not sufficiently controlled on inhaled steroid.

Altogether 170 patients, randomized to two treatment groups will be included. Key outcome measures are patient reported parameters on their asthma

DETAILED DESCRIPTION:
A phase IIb study in patients to evaluate CYT003- QbG10 versus placebo, in patients with mild to moderate allergic asthma not sufficiently controlled on inhaled steroid.

Altogether 170 patients, randomized to two treatment groups will be included. Key outcome measures are patient reported parameters on their asthma at the time of primary endpoint and throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Complete all protocol requirements.
3. Between 18 to 65 years of age.
4. Persistent allergic asthma patients
5. Forced expiratory volume in one second (FEV1) ≥60% to ≤ 90% of predicted value
6. Reversibility of airway obstruction
7. Patients meeting the contraception requirements
8. At baseline: Patients treated with ICS and insufficiently controlled
9. Blood eosinophil count above a certain level

Exclusion Criteria:

1. Failure to meet at least 80% compliance of use of the patient e-diary/ peak expiratory flow (PEF) meter (AM3 device) at the baseline visit
2. Treatment or hospitalization for asthma exacerbation within past 2 months
3. Current use or use of systemic corticosteroids within past 2 months
4. Current smokers.
5. Ex-smokers for less than 1 year, with a tobacco smoking history of >10 pack years
6. Major surgery within 3 months prior to signing the ICF or anticipated during study
7. Presence or history of clinically relevant cardiovascular, renal, pulmonary (e.g. COPD), endocrine, autoimmune, dermatological, neurological, psychiatric, or ocular disease as judged by the investigator.
8. Any malignancy within the previous 5 years
9. Presence of suspicious lymphadenopathy or splenomegaly on physical examination.
10. Confirmed or suspected current infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
11. Presence of active infectious disease as judged by the investigator
12. Active autoimmune diseases or prior diagnosis of autoimmune disease including but not limited to rheumatoid arthritis, lupus and ulcerative colitis.
13. Pregnancy (based on positive urine test at screening visit) or lactation.
14. Female planning to become pregnant during the study period.
15. Patients with any history of abuse of alcohol or other recreational drugs.
16. Ongoing or planned specific immunotherapy (SIT) during the whole study period or SIT completed within the last 3 years.
17. BMI >40
18. Use of investigational or approved biologics/immune-modulators within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Casale, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States